CLINICAL TRIAL: NCT02380170
Title: Epidemiology and Outcomes of Gram Negative Urosepsis
Acronym: SERPENS
Status: Completed | Type: Observational
Sponsor: European Association of Urology Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-01
Record Dates: First submitted 2014-11-20; First posted 2015-03-05 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Urosepsis
Keywords: sepsis; urinary tract infection; resistance; pathogens; mortality; health economics
MeSH Terms: conditions — Sepsis; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Urosepsis: Sepsis derived from the urinary tract infection

SUMMARY:
The study aims to get an insight on the causative bacteria of sepsis derived from the urinary tract. Furthermore, it is the intention to understand the outcomes of these patients. For this purpose a non-interventional, observational study will be conducted.

DETAILED DESCRIPTION:
In this prospective, non-interventional, observational registry participants diagnosed with urosepsis will be registered to the study to capture the events and outcomes of interest. There will be no additional intervention and evaluation for the purpose of this study.

-Primary objectives:

1. Pathogens: Causative pathogens and their susceptibility profile
2. Clinical outcomes: Development of organ failure and mortality.
3. Costs: Hospital resources used and costs acquired

   * Secondary objective:

<!-- -->

1. Risk factors: Influence of patient characteristics (medical & urological history, comorbidities) on severity of urosepsis (simple, severe & septic shock), causative pathogens profile and outcomes
2. Appropriateness of antibiotic treatment: The influence of appropriate antibiotic treatment, identified through empirical treatment provided and the pre-treatment culture results, on the clinical outcomes.
3. Economic evaluation: Identify the cost and health state changes according to appropriateness of treatment.

   -Rationale: Results of the GPIU registries 2003 to 2013 showed, that the rate of urosepsis in "health-care" associated infections of urological patients increased from 15% in 2003 to 25% in 2013. This creates an extra burden of health systems that needs to be better understood in detail.

   Early management in urosepsis is imperative. An important step of the management is appropriate empirical antibiotic treatment that requires an understanding of local and global pathogen susceptibility profiles. Furthermore, our pilot analysis from GPIU has shown that individual patient characteristics can be helpful in guiding empirical treatment. Appropriate empirical antibiotic treatment has shown to be associated with better clinical outcomes and lower length of stay (LOS).

   -Objectives

   The aim of this registry is to investigate the epidemiology of urosepsis primarily in Europe, with specific examination of causative pathogens and their resistance, the associated risk factors, clinical data, costs associated and value of initial appropriate antimicrobial treatment.

   3.1. Primary objectives:

   - Describe the prevalence of organisms causing urosepsis

   - Describe the susceptibility profile of organisms causing urosepsis.

   - Describe the clinical and economic burden of urosepsis caused by resistant Gram negative pathogens of interest.

   3.2. Secondary objectives:
   * Characterize risk factors for infection with resistant gram negative pathogens of interest.
   * Examine the impact of initial inappropriate antibiotic therapy on clinical and economic outcomes.
   * Design

   This is a prospective, longitudinal data collection as an ancillary registry to the 2013 Global Prevalence of Infections in Urology (GPIU) point prevalence registry performed annually by the European Association of Urology (European Section of Infection in Urology). Participating hospitals will perform data collection with a goal of collecting complete hospital course data on 600 cases of urosepsis. The GPIU group will handle contracting, data collection, and data analysis for this part of the registry.

   - Participants

   The population to be observed will be adults patients with clinical diagnosis of urosepsis. Observations will be initiated when a patient is diagnosed with urosepsis based on the clinical symptoms and findings as part of routine clinic practice through emergency and accident, urology or internal medicine units.

   The data of the bacterial isolates and their susceptibility results used in this study will be obtained as part of routine clinical care. The necessity of informed patient consent is at the discretion of the participating institution. All patient data will be analyzed anonymously.

   -Patients to be observed

   Identification of observations:

   Patients to be observed will be identified through emergency and accident, urology, intensive care and internal medicine units at participating sites. Eligibility criteria checklist of all cases considered to be observed will be filled in by participating principal investigator (PI). Clinical information from the initial diagnosis should be used to asses eligibility.

   -Observations Diagnosis observations

   Routine clinical signs and symptoms assessed by the managing physician should be used to evaluate the patient. The following observations should be carried out at the time of diagnosis:
   * Medical history
   * Microbiology cultures
   * Clinical signs, symptoms and findings

   Treatment observations

   The following observations should be registered after the diagnosis and initiation of treatment:
   * Medical treatment
   * Surgical treatment
   * Treatment unit

   Post-treatment observations

   Subsequent to initiation of treatment the following observations will be registered:

   • End organ failure
   * Shift in treatments
   * Mortality

   Registration will be carried out on post diagnosis day 3,7,9 and 30 to capture the changes within the following time-gaps respectively:
   * Diagnosis day to day 3
   * Post diagnosis day 4 to 7
   * Post diagnosis day 8 to 9
   * Post diagnosis day 10 to 30

   For patients where treatment extends beyond 30 days additional registrations will be carried out only when there is a change in the listed post-treatment observations.

   Completion of treatment - observations

   When treatment of patients is finalized due to either complete resolution of sepsis or death the following observations will be carried out:

   • Costs (optional)
   * End-organ failure
   * Mortality
   * LOS
   * HRQoL (optional)

   Post diagnosis 1 year follow-up

   At the end of 1st year of diagnosis centers willing to register further observations will fill in the following:

   • Costs (optional)

   • End-organ failure

   • Mortality

   • LOS

   • HRQoL (optional)

   Schedule of observations

   - Baseline: Medical history, Microbiological proof, management of urosepsis, HRQoL(optional)

   -Follow-up-1 (3rd day post diagnosis): Microbiological proof(if additional carried out), Management of urosepsis, Clinical outcomes

   -Follow-up-2 (7th day post diagnosis): Microbiological proof(if additional carried out), Management of urosepsis, Clinical outcomes
   * Follow-up-3 (9th day post diagnosis): Microbiological proof(if additional carried out), Management of urosepsis, Clinical outcomes
   * Follow-up-4 (30th day post diagnosis): Microbiological proof(if additional carried out), Management of urosepsis, Clinical outcomes
   * Completion of treatment related with urosepsis episode: Management of urosepsis, Clinical outcomes, HRQoL (optional), Economic evaluation (optional)
   * Statistical considerations Data measured on a continuous scale will be expressed as mean, standard deviation, range, and median. Categorical data will be expressed as counts and percentages of patients in the categories. Chi-square or Fisher's tests will be used to test for statistical differences in categorical variables and T- or Mann-Whitney tests will be utilized for determination of statistical differences in continuous variables where appropriate.
   * Management The GPIU study team will provide support for the participating centers. The secretarial staff at the EAU-Research foundation will provide clerical support to the study.
   * Administration, logistics & quality assurance

   Sharing of observations

   Electronic (e) case report forms (CRF) will be used for collection of observational information. EAU-RF will and study coordinator will provide guidance to sites to aid the completion of the eCRFs. The study scientific group reserves the right to amend or add to the eCRF template as appropriate. Such changes to not constitute a protocol amendment and revised or additional forms should be used by sites.

   Central data monitoring:

   After eCRFs are completed by the study site, the study coordinator will review it for protocol compliance, and for inconsistencies and missing values.

   Should any missing data or data abnormalities be found, queries will be raised for resolution by the site.

   Any systematic inconsistencies identified through central data monitoring may be subject to queries.

   Definition of end of registry:

   The end of the study will be the date of the last observation captured.

ELIGIBILITY:
Inclusion Criteria:

* Microbiologically proven UTI
* Age>18
* Patients must meet at least two of the following four SIRS criteria, at least one of which must be the core temperature criterion or the WBC criterion; these criteria did not have to be met simultaneously:

  1. Hypothermia by core temperature <36ºC, or hyperthermia >38ºC measured via any means
  2. Heart rate (HR) >90 beats per minute
  3. Respiratory rate (RR) >20 breaths/minute related to septic event, or partial pressure of arterial carbon dioxide (PaCO2) <32 mmHg related to septic event or requiring mechanical ventilation related to septic event
  4. Total WBC absolute count >12,000 cells/mm3 presence of granulocyte-stimulating factor, for those patients whose WBC absolute count was >12,000 cells/mm3 one other criterion (RR or HR) or <4000 cells/mm3. In the , they must have had a fever and at least

Exclusion Criteria:

* Sepsis due to other causes besides the urogenital tract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population to be observed will be adults patients with clinical diagnosis of urosepsis. Observations will be inititated when a patient is diagnosed with urosepsis based on the clinical symptoms and findings as part of routine clinic practice through emergency and accident, urology or internal medicine units.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-08-24 (Actual); Study Completion 2020-05-24 (Actual)

PRIMARY OUTCOMES:
Number of patients with each causative pathogens and their susceptibility profile at the baseline evaluation (diagnosis of urosepsis) | initial diagnosis of urosepsis
  Analysis results of microbiological cultures will be used to group them according to the definitions suggested by the ECDC as multi-drug resistant (MDR), extensive drug resistant (XDR) and pan-drug resistant (PDR).

SECONDARY OUTCOMES:
Hospital Costs (Euros) of each patients Urosepsis management | Duration of Hospitalisation (basline evaluation to discharge of patient or death)
All cause mortality | First 30 days from diagnosis
  Mortality will be captured and the reason of death will also be recorded
Morbidity | First 30 days from diagnosis (baseline)
  Development of organ failure i. Kidney failure ii. Cardiovascular failure iii. Pulmonary failure iv. Hepatic failure v. Ileus vi. Thrombocytopenia
Health related Quality of Life | Baseline, Follow-up (3rd, 7th, 9th and 30th day after baseline)
  EQ-5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Truls Erik Bjerklund Johansen, Prof., Study Chair — Oslo Univeristy, Norway; Florian Wagenlehner, Prof., Study Chair — Giessen Univeristy, Germany; Zafer Tandogdu, MD, Study Director — Northern Institute for Cancer Research, Newcastle University, UK
Locations (7):
- South-Pest Teaching Hospital, Budapest, Hungary
- Manzoni Hospital, Lecco, Italy
- University Clinic of Surgery " St. Naum Ohridski", Skopje, North Macedonia
- Oslo University Hospital, Oslo, Norway
- Nicolaus Copernicus City Hospital, Torun, Poland
- Centro Hospitalar Cova da Beira, Lisbon, Portugal
- GOP Taksim Teaching Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Angus DC, Wax RS. Epidemiology of sepsis: an update. Crit Care Med. 2001 Jul;29(7 Suppl):S109-16. doi: 10.1097/00003246-200107001-00035. PMID 11445744
- [Background] Tandogdu Z, Cek M, Wagenlehner F, Naber K, Tenke P, van Ostrum E, Johansen TB. Resistance patterns of nosocomial urinary tract infections in urology departments: 8-year results of the global prevalence of infections in urology study. World J Urol. 2014 Jun;32(3):791-801. doi: 10.1007/s00345-013-1154-8. Epub 2013 Aug 24. PMID 23979151
- [Derived] Tandogdu Z, Koves B, Ristovski S, Balci MBC, Rennesund K, Gravas S, Nale D, Medina-Polo J, Garabasova MK, Costantini E, Cano-Valasco J, Glavinova MS, Bruyere F, Perepanova T, Kulchavenya E, Cek M, Wagenlehner F, Johansen TEB; SERPENS Investigators. Urosepsis 30-day mortality, morbidity, and their risk factors: SERPENS study, a prospective, observational multi-center study. World J Urol. 2024 May 10;42(1):314. doi: 10.1007/s00345-024-04979-2. PMID 38730089
- See also: Study webpage — https://gpiu-serpens.org/